CLINICAL TRIAL: NCT00466934
Title: Cross-Validating NIRS With fMRI
Brief Title: Measuring Blood Flow in the Brain
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: United States Department of Defense (U.S. Federal Agency); National Institutes of Health Clinical Center (CC) (NIH); Center for Neuroscience and Regenerative Medicine (CNRM) (U.S. Federal Agency)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070139; 07-N-0139
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-12-29

CONDITIONS: Traumatic Brain Injury; Healthy
Keywords: Cerebral Blood Flow; Cerebral Cortex; Cognition; Optical Imaging; Healthy Volunteer; HV
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will test a method of measuring brain blood flow called near infrared spectroscopy (NIRS). It will determine whether NIRS gives the same results as the more commonly used technique, functional magnetic resonance imaging (fMRI).

Healthy normal volunteers between 18 and 60 years of age may be eligible for this study. Participants come to the NIH up to six times for experiments using NIRS and fMRI. They do the following tasks while they are undergoing NIRS or fMRI:

* looking at a computer monitor while a checkerboard pattern changes
* wiggling the toes and moving the fingers
* Reading words on a computer screen and pushing one button if they are plants and another if they are animals.

For NIRS, a frame is placed on the head and held it in place with a metal band. The frame holds sensors that contact the scalp.

For fMRI, the subject lies on a table that can slide in and out of an MRI scanner, a metal cylinder surrounded by a strong magnetic field. fMRI uses a strong magnetic field and radio waves to obtain images of the brain while the subject performs tasks. During the procedure, The subject wears earplugs to muffle the sound of loud knocking noises that occur during scanning.

DETAILED DESCRIPTION:
OBJECTIVE: a) to explore the usefulness of Near Infrared Spectroscopy (NIRS) as a means of mapping brain activity, to see whether the results are similar to those of fMRI and b) to see whether spontaneous brain blood flow changes coincide with changes in behavior.

STUDY POPULATION: 50 healthy volunteers.

DESIGN: The study will look for correlations between NIRS and fMRI signal changes in the same subjects. It will also detect relationships between spontaneous blood flow shifts and shifts and changes in cognitive performance. Finally, NIRS will be combined with a frontal lobe activation task to see if blood flow changes can be detected over the hairless skin of the forehead in a simple, standardized manner that might yield a diagnostic test for frontal injury.

OUTCOME MEASURES: Graded changes in blood flow and oxygen, measured with NIRS and fMRI and variations in response time on a word task.

ELIGIBILITY:
* INCLUSION CRITERIA:

Age 18 to 60, inclusive.

EXCLUSION CRITERIA:

* Pregnancy.
* History of hypertension.
* History of any disease of the central nervous system.
* Current use of sedating medication, including antihistamines.
* Subjects with any of the following will be excluded from MRI testing: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or auto-defibrillator; cochlear implant; ocular foreign body, such as metal shavings; permanent eyeliner; insulin pump; or irremovable body piercing due to the possible dangerous effects of the MRI magnet upon metal objects in the body.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2007-04-24; Study Completion 2011-12-29

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Benaron DA, Hintz SR, Villringer A, Boas D, Kleinschmidt A, Frahm J, Hirth C, Obrig H, van Houten JC, Kermit EL, Cheong WF, Stevenson DK. Noninvasive functional imaging of human brain using light. J Cereb Blood Flow Metab. 2000 Mar;20(3):469-77. doi: 10.1097/00004647-200003000-00005. PMID 10724111
- [Background] Biswal B, Hudetz AG, Yetkin FZ, Haughton VM, Hyde JS. Hypercapnia reversibly suppresses low-frequency fluctuations in the human motor cortex during rest using echo-planar MRI. J Cereb Blood Flow Metab. 1997 Mar;17(3):301-8. doi: 10.1097/00004647-199703000-00007. PMID 9119903
- [Background] Biswal B, Yetkin FZ, Haughton VM, Hyde JS. Functional connectivity in the motor cortex of resting human brain using echo-planar MRI. Magn Reson Med. 1995 Oct;34(4):537-41. doi: 10.1002/mrm.1910340409. PMID 8524021